CLINICAL TRIAL: NCT02392416
Title: Non-interventional, Multicenter Clinical Study to Assess the Treatment With Atorvastatin in Patient Compliance With Hyperlipidemia and Other Cardiovascular Risk Factors
Brief Title: Atorvastatin Study in Cardiovascular Disease Risk
Acronym: ANTLER
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-ATR-EL-56
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Hypercholesterolemia; Dyslipidemia
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Treatment of hypercholesterolemia is based on the guidelines of ESC-EAS 2011 (European Heart Journal (2011) 32, 1769-1818, ESC / EAS Guidelines for the management of dyslipidaemias) These calculate the 10 year risk based on SCORE tables - Systematic COronary Risk Estimation and taking into account specific parameters in the patient's profile.

DETAILED DESCRIPTION:
The European Society of Cardiology initiated the development of a new risk calculation system (SCORE) using data from 12 European population monitoring studies (N = 205.178) with wide geographic distribution of countries with different cardiovascular risk. The SCORE data contains more than 3 million man-years of observation and 7934 fatal cardiovascular events.

* patient is classified into risk category (Very high-high-medium-low)
* a target for LDL-C was then placed on a risk basis and appropriate treatment proposed
* As a first option is to statin monotherapy to the maximum tolerated dose.
* Only in case of failure of the therapeutic target for LDL-C may be used active substance other therapeutic class or as alternative monotherapy or in combination with statin, Because European countries exhibit heterogeneity in genetics, lifestyle, living standards, health benefits, etc. have been divided into two groups, high risk (countries) and low risk (countries) and have been prepared in different tables SCORE (Systematic COronary Risk Estimation) For Greece, as in other countries has been further refinement of SCORE and trained specialists tables adapted to the Greek population (Statistical The most currently used treatment in Greece is atorvastatin, obtained from 520,000 patients From far studies with atorvastatin have been well documented reductions in various lipid parameters and especially the LDL-C, which is the main objective in the treatment.

But there is no evidence to suggest what is the dosage proved suitable in practice for the patient depending on the risk class belongs.

ELIGIBILITY:
Inclusion Criteria:

* External outpatients who monitored externally hospital lipid clinic, hypercholesterolemia, diabetic etc.
* Male or female
* Eligible ages for the study: 18-99 years
* Patients with a first diagnosis of hypercholesterolemia who are to receive Atorvastatini according to standard clinical practice
* Established cardiovascular disease by interventional or non-interventional examinations (such as coronary angiography, nuclear medicine, echocardiography stress, carotid plaque ultrasound), previous myocardial infarction, ACS, coronary revascularization (PCI, CABG), and other arterial revascularization procedures, ischemic stroke, peripheral arterial disease (PAD)
* Diabetes mellitus (type 1 or type 2) with one or more cardiovascular risk factors and / or target organ damage (such as microalbuminuria: 30-300 mg / 24 h)
* Patients already diagnosed with hypercholesterolemia and unregulated who will receive Atorvastatini according to standard clinical practice
* Patients diagnosed and set to original formulation of atorvastatin
* Patients who have fully understood the study protocol and signed the consent form

Exclusion Criteria:

* Patients <18 years
* Hypersensitivity to atorvastatin or to any of the excipients
* Women pregnant or breastfeeding
* Patients who have not fully understood the study protocol and have not signed the consent form

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dyslipidemia
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
SCORE - Systematic COronary Risk Estimation | 4 months
  Estimation of SCORE

SECONDARY OUTCOMES:
Compliance (Change in 8-item Morisky Scale) | 4 months
  Change in 8-item Morisky Scale

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Gennimatas General State Hospital, Athens, Attica
  - 2nd Cardiology Department,, University of Athens, Attikon Hospital, Haidari, Athens

REFERENCES:
- [Background] Pitsavos C, Panagiotakos DB, Chrysohoou C, Stefanadis C. Epidemiology of cardiovascular risk factors in Greece: aims, design and baseline characteristics of the ATTICA study. BMC Public Health. 2003 Oct 20;3:32. doi: 10.1186/1471-2458-3-32. PMID 14567760
- [Background] Panagiotakos DB, Pitsavos C, Manios Y, Polychronopoulos E, Chrysohoou CA, Stefanadis C. Socio-economic status in relation to risk factors associated with cardiovascular disease, in healthy individuals from the ATTICA study. Eur J Cardiovasc Prev Rehabil. 2005 Feb;12(1):68-74. PMID 15703509
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Krousel-Wood M, Islam T, Webber LS, Re RN, Morisky DE, Muntner P. New medication adherence scale versus pharmacy fill rates in seniors with hypertension. Am J Manag Care. 2009 Jan;15(1):59-66. PMID 19146365
- [Result] Morisky DE, DiMatteo MR. Improving the measurement of self-reported medication nonadherence: response to authors. J Clin Epidemiol. 2011 Mar;64(3):255-7; discussion 258-63. doi: 10.1016/j.jclinepi.2010.09.002. Epub 2010 Dec 8. No abstract available. PMID 21144706